CLINICAL TRIAL: NCT00815867
Title: Effect of Epoetin Beta on Renal Function Within 30 Days Following a Kidney Transplant
Acronym: Neo-PDGF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI07-PR-CHOUKROUN; 2007/14 CPP; 2007-002562-35 EudraCT
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Kidney Failure
Keywords: kidney failure; kidney transplant; graft function; haemoglobin; epoetin
MeSH Terms: conditions — Renal Insufficiency | interventions — epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patient will receive Epoetin Beta
  Interventions: Drug: epoetin beta (NeoRecormon ®)
- B (No Intervention)

INTERVENTIONS:
Drug: epoetin beta (NeoRecormon ®) — comparison of administration of high dosage of epoetin vs no administration of epoetin
  30000 UI: 4 injections
  Other Names: Neorecormon
  Arms: A

SUMMARY:
Main objective : Assessing the effect of epoetin beta on Hb rate and the glomerular filtration rate estimated 30 days after kidney transplant.

DETAILED DESCRIPTION:
French study, prospective, multicenter, open, randomized into two parallel groups:

Group A: NeoRecormon ® 30000 UI: 4 injections Group B: control group without administration of the medical product

Period of recruitment: 18 months Duration of participation of each patient: 90 days Total duration of the test: 21 months.

Main objective : Assessing the effect of epoetin beta on the glomerular filtration rate estimated 30 days after kidney transplant.

Secondary objectives:

Comparing the 2 groups at all times J0 to J90:

* The evolution of renal function
* The survival of patients and grafts
* The time of onset and incidence of acute rejection proved by biopsy
* The correction of anemia
* The need for transfusions
* The need for EPO
* Quality of Life
* The safety processing

ELIGIBILITY:
Inclusion Criteria:

* Males anf Females aged between 18 and 75
* Patients having given their written consent
* Patient determined to participate in the test and to respect the requirements
* Patient covered by a social insurance
* Patient to be kidney transplanted (from a cadaveric donor)
* Patient benefiting from the 1st or 2nd kidney transplant
* Patient formerly treated by peritoneal dialysis or hemodialysis
* Patient receiving a graft with risk of delayed graft function (score> 7 combining age of the donor, ischemia time, receiver ethnicity and cause of death)
* Patient to receive treatment with basiliximab, mycophenolate mofetil, tacrolimus and corticosteroid

Exclusion Criteria:

* Patient Pregnant or nursing
* Patient with a disability that does not ensure the good understanding of the study and its imperatives , or patient having dependency (alcohol, drugs)
* Patient receiving doses of epoetin beta or alpha> 30,000 IU / week or darbepoetin> 150 microg / week before transplanting
* Patient who has participated in a clinical trial in the last month or currently included in another test
* Patient in safeguarding justice, guardianship or trusteeship
* Patient receiving a third transplant or hyper immune or who have a positive historic cross-match
* Patient receiving a preemptive transplant
* graft from a living donor
* graft with 3 or more arteries
* Multi-Organ Transplantation
* Patient with heart failure stage> III
* Patients with unstable ischemic heart disease, or have had a major coronary event less than 6 months, stroke or TIA <6 months or symptomatic arteritis of lower limbs stage ≥ 3
* Patients with active viral infection: hepatitis B, C (PCR + only) or HIV
* Patient with a history of anemia from erythroblastopenia
* Patient receiving anticoagulant treatment(AVK) before renal transplantation and to be continued after transplant
* Patient with a preoperative rate Hb> 14 g / dL (before ultrafiltration)
* A patient with known hypersensitivity to the active substance or to any of the excipients, or to benzoic acid
* Patients with poorly controlled hypertension in the weeks before transplantation (Diastolic Blood Pressure ≥ 110 mm Hg with more than 3 antihypertensive drugs)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Assessing the effect of epoetin beta on the glomerular filtration rate estimated 30 days after kidney transplant | 30 days

SECONDARY OUTCOMES:
The evolution of renal function | 90 days
The survival of patients and grafts | 90 days
The time of onset and incidence of acute rejection proved by biopsy | 90 days
The correction of anemia | 90 days
The need for transfusions | 90 days
The need for EPO | 90 days
Quality of Life | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: CHOUKROUN Gabriel, Ph D, Principal Investigator — CHU Amiens; MARTINEZ Franck, Ph D, Principal Investigator — Necker Hospital
Locations (17):
- France (17):
  - Amiens hospital, Amiens
  - LA CAVALE BLANCHE Hospital, Brest
  - MONDOR Hospital, Créteil
  - MICHALLON Hospital, Grenoble
  - Kremlin Bicêtre Hospital, Le Kremlin-Bicêtre
  - ALBERT CALMETTE Hospital, Lille
  - CHU Nantes, Hotel-Dieu Hospital, Nantes
  - CHU Nice, Pasteur Hospital, Nice
  - Georges Pompidou European Hospital, Paris
  - TENON Hospital, Paris
  - Necker Hospital, Paris
  - LA MILETRIE Hospital, Poitiers
  - MAISON BLANCHE Hospital, Reims
  - Bois Guillaume Hospital, Rouen
  - FOCH Hospital, Suresnes
  - RANGUEIL Hospital, Toulouse
  - BRETONNEAU Hospital, Tours

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Martinez F, Kamar N, Pallet N, Lang P, Durrbach A, Lebranchu Y, Adem A, Barbier S, Cassuto-Viguier E, Glowaki F, Le Meur Y, Rostaing L, Legendre C, Hermine O, Choukroun G; NeoPDGF Study Investigators. High dose epoetin beta in the first weeks following renal transplantation and delayed graft function: Results of the Neo-PDGF Study. Am J Transplant. 2010 Jul;10(7):1695-700. doi: 10.1111/j.1600-6143.2010.03142.x. PMID 20642691